CLINICAL TRIAL: NCT01436162
Title: The SPD489-323 Phase 3, Multicenter, Randomized, Double-blind, Parallel-group, Placebo-controlled, Flexible Dose Titration, Efficacy and Safety Study of SPD489 in Combination With an Antidepressant in the Treatment of Adults With Major Depressive Disorder With Inadequate Response to Prospective Treatment With an Antidepressant
Brief Title: Efficacy and Safety Study of SPD489 in Combination With an Antidepressant in the Treatment of Adults With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPD489-323; 2011-003006-25 (EudraCT Number)
Record Dates: First submitted 2011-09-15; First posted 2011-09-19 (Estimated); Results first posted 2014-11-07 (Estimated); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Antidepressive Agents; Lisdexamfetamine Dimesylate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Antidepressant + SPD489 (Experimental)
  Interventions: Drug: Antidepressant + SPD489 (Lisdexamfetamine dimesylate )
- Antidepressant + Placebo (Placebo Comparator)
  Interventions: Drug: Antidepressant + Placebo

INTERVENTIONS:
Drug: Antidepressant + SPD489 (Lisdexamfetamine dimesylate ) — Antidepressant (either escitalopram oxalate, sertraline hydrochloride, venlafaxine hydrochloride extended release or duloxetine hydrochloride) oral, once daily + SPD489 (oral, 20, 30, 50 or 70 mg, once daily) for 8 weeks
  Other Names: Vyvanse
  Arms: Antidepressant + SPD489
Drug: Antidepressant + Placebo — Antidepressant (either escitalopram oxalate, sertraline hydrochloride, venlafaxine hydrochloride extended release or duloxetine hydrochloride) oral, once daily + Placebo (oral, once daily) for 8 weeks
  Arms: Antidepressant + Placebo

SUMMARY:
This study will examine SPD489 in subjects aged 18-65 with major depressive disorder (MDD) who are taking certain types of antidepressants but continue to have residual depression symptoms. Eligible patients will remain on their antidepressant but will be randomized to either receive supplemental SPD489 or placebo (i.e. sugar pill). The purpose of this study is to help answer the following questions:

* How safe is SPD489 for the supplemental treatment of depression and what are the side effects that might be related to it?
* Can supplemental SPD489 help patients who still have residual depression symptoms while taking an antidepressant?
* How much SPD489 should be given to patients with depression who are also taking an antidepressant?
* How does SPD489 compare to placebo in depressed patients who are also taking an antidepressant?

ELIGIBILITY:
Inclusion Criteria

1. Subject is able to provide written, personally signed, and dated informed consent to participate in the study before completing any study-related procedures.
2. Subject is between 18 and 65 years of age.
3. Subject has a primary diagnosis of non-psychotic MDD.
4. Subject has a MADRS total score >/=24.
5. Subject is willing and has an understanding and ability to fully comply with study procedures and restrictions defined in this protocol.
6. Subject, who is female, must have a negative serum beta human chorionic gonadotropin (B-HCG) pregnancy test and a negative urine pregnancy test and agrees to comply with any applicable contraceptive requirements of the protocol.
7. Subject is able to swallow a capsule.

Exclusion Criteria:

1. Subject whose current episode of MDD has not responded to an adequate treatment regimen with 2 or more approved single antidepressant agents.
2. Subject who has a lifetime history of treatment resistant depression, defined as having not responded to adequate treatment with 2 or more treatment regimens.
3. Subject has a current co-morbid psychiatric disorder that is either controlled with medications prohibited in this study or is uncontrolled and associated with significant symptoms.
4. Subject has been hospitalized (within the last 12 months) for their current MDD episode.
5. Subject has a current or lifetime history of attention-deficit/hyperactivity disorder (ADHD).
6. Subject has a first degree relative that has been diagnosed with bipolar I disorder.
7. Subject has a recent history (within the last 6 months) of suspected substance abuse or dependence disorder.
8. Subject is considered a suicide risk, has previously made a suicide attempt within the past 3 years, or is currently demonstrating active suicidal ideation.
9. Subject has a concurrent chronic or acute illness or unstable medical condition.
10. Subject has a history of seizures (other than infantile febrile seizures), any tic disorder, or a current diagnosis and/or a known family history of Tourette's Disorder, serious neurological disease, history of significant head trauma, dementia, cerebrovascular disease, Parkinson's disease, or intracranial lesions.
11. Subject has known history of symptomatic cardiovascular disease, advanced arteriosclerosis, structural cardiac abnormality, cardiomyopathy, serious heart rhythm abnormalities, coronary artery disease, or other serious cardiac problems.
12. Subject has a history of thyroid disorder that has not been stabilized on thyroid medication or treatment within 3 months prior to the Screening Visit.
13. Subject has a known family history of sudden cardiac death or ventricular arrhythmia.
14. Subject has glaucoma.
15. Subject has any clinically significant ECG or clinical laboratory abnormalities.
16. Subject has a history of moderate to severe hypertension.
17. Current use of any other medications (including over-the-counter [OTC], herbal or homeopathic preparations) that have central nervous system effects.
18. Subject has the potential need to initiate or modify frequency of psychotherapy or to continue or initiate other treatments for depression, outside of those allowed in this protocol.
19. Subject has had electroconvulsive therapy (ECT) for the current depressive episode 3 months prior to the Lead-in Baseline Visit.
20. The subject has a known or suspected intolerance or hypersensitivity to the investigational product.
21. The subject has a known or suspected intolerance, hypersensitivity, or contraindications to their assigned antidepressant treatments (escitalopram oxalate, sertraline HCl, venlafaxine HCl extended release, or duloxetine HCl).
22. Subject has a positive urine drug result.
23. Subject has a body mass index (BMI) of <18.5 or >40.
24. Subject is female and is pregnant or nursing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1105 (Actual)
Dates: Start 2011-10-19 (Actual); Primary Completion 2013-12-10 (Actual); Study Completion 2013-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (101):
- United States (36):
  - ResearchOne, Inc., Scottsdale, Arizona
  - K&S Professional Research Services, LLC, Little Rock, Arkansas
  - ATP Clinical Research, Inc., Costa Mesa, California
  - Diligent Clinical Trials, Downey, California
  - Synergy Clinical Reserach Center of Escondido, Escondido, California
  - Pacific Research Partners, LLC, Oakland, California
  - Anderson Clinical Research, Redlands, California
  - BreakThrough Clinical Trials, LLC, San Bernardino, California
  - MCB Clinical Research Centers, Colorado Springs, Colorado
  - Florida Clinical Research Center, LLC, Bradenton, Florida
  - Scientific Clinical Research, Inc., North Miami, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Comprehensive NeuroScience, Inc., St. Petersburg, Florida
  - Janus Center for Psychiatric Research, West Palm Beach, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Atlanta Institute of Medicine & Research, Atlanta, Georgia
  - Pedia Research, Newburgh, Indiana
  - Heartland Research Associates, Wichita, Kansas
  - Louisiana Clinical Research, LLC, Shreveport, Louisiana
  - Comprehensive Psychiatric Associates, Gladstone, Missouri
  - The Center for Pharmaceutical Research, Kansas City, Missouri
  - Mercy Health Research, St Louis, Missouri
  - Bio Behavioral Health, Toms River, New Jersey
  - Brooklyn Medical Institute, Brooklyn, New York
  - Medical & Behavioral Health Research, PC, New York, New York
  - Midwest Clinical Research Center, Dayton, Ohio
  - North Star Medical Research, LLC, Middleburg Heights, Ohio
  - Sooner Clinical Research, Oklahoma City, Oklahoma
  - Lehigh Center for Clinical Research, Allentown, Pennsylvania
  - Belmont Center for Comprehensive Treatment, Philadelphia, Pennsylvania
  - Medical University South Carolina Anxiety Disorder Program, North Charleston, South Carolina
  - Psychiatric Consultants, PC, Franklin, Tennessee
  - Research Strategies of Memphis, LLC, Memphis, Tennessee
  - KRK Medical Research, Dallas, Texas
  - Future Search Trials of Dallas, LP, Dallas, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
- Dr Lieven De Weirdt, Sint-Niklaas, Belgium
- Czechia (9):
  - Saint Anne s.r.o., Brno
  - Psychiatricka ambulance, Brno
  - Medicana s.r.o., Hořovice
  - Psychiatrie s.r.o., Kutná Hora
  - Bialbi s.r.o., Litoměřice
  - Clintrial s.r.o., Prague
  - Psychiatry Trial s.r.o., Prague
  - Prague Medical Services s.r.o., Prague
  - Ricany s.r.o., Říčany
- Estonia (5):
  - Parnu Hospital, Psychiatric Clinic, Pärnu
  - North Estonia Medical Centre Foundation Psychiatry Clinic, Tallinn
  - Marienthal Psychiatry and Psychology Center, Tallinn
  - Jaanson & Laane OU, Tartu
  - Tartu University Hospital Psychiatric Clinic, Tartu
- Finland (4):
  - ARTES Psykiatrinen Palvelukeskus Oy, Helsinki
  - Satucon Oy, Kuopio
  - Satakunnan Psykiatripalveiu Oy at Mentoria Oy, Tampere
  - Puutorin Psykiatripalvelu, Turku
- Germany (14):
  - Gemeinschafstpraxis für Neurologie und Psychiatrie, Psychotherapie, Achim
  - Private Praxis Dr. Jana Thomsen, Berlin
  - emovis GmbH, Berlin
  - Alexander Schulze, MD, Berlin
  - Private Practice Drs. Bitter/Schumann, Bochum
  - University Hospital Carl Gustav Carus, Dresden
  - ZSL Zentrum fuer medizinische Studien in Leipzig, Leipzig
  - Studienzentrum Muenchen, München
  - Universitaetsklinikum Munster, Münster
  - Studienzentrum Klinikum Nuernberg, Nuremberg
  - Somni bene GmbH, Schwerin
  - Private Practice: Eugen Schlegel, Siegen
  - Studiezentrum Nord-West, Westerstede
  - Medizinisches Studienzentrum Wuerzburg, Würzburg
- Hungary (5):
  - Semmelweis Univ. Dept.of Psychiatry, Budapest
  - Debrecent Egyetem Orvos es Egeszsegtudomanyl Centrum Pszichiatrai, Debrecen
  - Santha Kalman Mentalis Egeszsegkozpont es Szakkorhaz, Nagykálló
  - Josa Andras Teaching Hospital, Nyíregyháza
  - Pecsi Tudomanyegyeiem Pszichiatriai es Pszichoterapias Klinika, Sziget
- Poland (9):
  - Prywatne Gabinety Lekarskie "Promedicus", Bialystok
  - NZOZ Centrum Kultury, Higieny i Zdrowia Psychicznego, Bydgoszcz
  - Zespol Opieki Zdrowotnej w Chelmnie, Chełmno
  - Centrum Badan Klinicznuch Pl-House sp. z.o.o., Gdansk
  - Klinika Chorob Psychicznych i Zaburzen Nerwicowych, Gdansk
  - Centrum Psychiatrii i Psychoterapli, Gorlice
  - NZOZ Syntonia, Poradnia Zdrowia Psychicznego, Kielce
  - Osrodek Badafi Klinicznych Prof dr hab n med Meszek Szczepanski Prywatna Praktyka Lekarska, Lublin
  - Samodzielny Publiczny Zespol Zakladow Opieki Zdrowotnej w Zurominie, Żuromin
- Romania (6):
  - Spitatul Clinic Judetean de Urgenta Arad, Clinica de Psihiatrie, Arad
  - Stefi-Dent SRL, Botoșani
  - Spitalui Clinic de Psihiatrie "Prof. Dr. Alexandru Obregia" Sectia Clinica Psihiatrie I, Bucharest
  - Crucea Alba, Oradea
  - Lorentina 2201 SRL, Târgovişte
  - Spitalul Clinic Judetean Mures, Târgu Mureş
- South Africa (6):
  - Cape Trial Centre, Bellville, Cape Town
  - Flexivest Fourteen Research Centre, Bellville, Cape Town
  - Private Practice - Gerta Brink, Johannesburg, Gauten
  - Somerset West Clinical Research, Somerset West, Western Cape
  - Vista Clinic, Centurion
  - George Medi Clinic Extension, George
- Sweden (6):
  - SU/ Affektiva 1, Gothenburg
  - ProbarE i Lund AB, Lund
  - Ekdahl Medical AB, Malmo
  - INM Psykiatrisk Mottagning, Malmo
  - Medinstructor Lippitz AB, Stockholm
  - Dr. Wahlstedts mottagning, Uppsala

REFERENCES:
- [Result] Richards C, McIntyre RS, Weisler R, Sambunaris A, Brawman-Mintzer O, Gao J, Geibel B, Dauphin M, Madhoo M. Lisdexamfetamine dimesylate augmentation for adults with major depressive disorder and inadequate response to antidepressant monotherapy: Results from 2 phase 3, multicenter, randomized, double-blind, placebo-controlled studies. J Affect Disord. 2016 Dec;206:151-160. doi: 10.1016/j.jad.2016.07.006. Epub 2016 Jul 5. PMID 27474961

RESULTS

PARTICIPANT FLOW:
Groups:
- Antidepressant + Single-blind Placebo: Subjects received unblinded oral, once daily standard antidepressant therapy (either escitalopram oxalate, sertraline hydrochloride, venlafaxine hydrochloride extended release, or duloxetine hydrochloride) plus oral, once daily placebo (matching SPD489).
- Antidepressant + Double-blind SPD489: Subjects received assigned oral, once daily antidepressant therapy (either escitalopram oxalate, sertraline hydrochloride, venlafaxine hydrochloride extended release, or duloxetine hydrochloride), plus oral, once daily SPD489 (Lisdexamfetamine dimesylate optimized among a 20, 30, 50, or 70 mg dose).
- Antidepressant + Double-blind Placebo: Subjects received assigned oral, once daily antidepressant therapy (either escitalopram oxalate, sertraline hydrochloride, venlafaxine hydrochloride extended release, or duloxetine hydrochloride) plus oral, once daily, double-blind placebo (matching SPD489).
Period: Single-blind Lead-in Phase
Arm/Group | Antidepressant + Single-blind Placebo | Antidepressant + Double-blind SPD489 | Antidepressant + Double-blind Placebo
Started | 1105 (Ten subjects were enrolled but not dosed.) | 0 | 0
Completed | 823 | 0 | 0
Not Completed | 282 | 0 | 0
Not completed — Adverse Event | 26 | 0 | 0
Not completed — Protocol Violation | 24 | 0 | 0
Not completed — Withdrawal by Subject | 69 | 0 | 0
Not completed — Lost to Follow-up | 43 | 0 | 0
Not completed — Met BP or Pulse Withdrawal Criteria | 13 | 0 | 0
Not completed — Other | 107 | 0 | 0
Period: Randomized Phase
Arm/Group | Antidepressant + Single-blind Placebo | Antidepressant + Double-blind SPD489 | Antidepressant + Double-blind Placebo
Started | 397 (These subjects were not included in the Safety Analysis Set or Full Analysis Set.) | 212 (One subject was randomized to this arm but did not receive at least 1 dose of double-blind treatment) | 214 (One subject was randomized to this arm but did not receive at least 1 dose of double-blind treatment)
Completed | 353 | 181 | 189
Not Completed | 44 | 31 | 25
Not completed — Adverse Event | 1 | 5 | 6
Not completed — Protocol Violation | 4 | 4 | 2
Not completed — Withdrawal by Subject | 16 | 9 | 8
Not completed — Lost to Follow-up | 17 | 5 | 4
Not completed — Lack of Efficacy | 0 | 1 | 1
Not completed — Met BP Or Pulse Withdrawal Criteria | 4 | 2 | 0
Not completed — Other | 2 | 5 | 4

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: All subjects who took at least 1 dose of randomized investigational product and who had at least 1 safety assessment.
Groups:
- Antidepressant + Double-blind SPD489: Subjects received assigned oral, once daily antidepressant therapy (either escitalopram oxalate, sertraline hydrochloride, venlafaxine hydrochloride extended release, or duloxetine hydrochloride), plus oral, once daily SPD489 (Lisdexamfetamine dimesylate optimized among a 20, 30, 50, or 70 mg dose) for 8 weeks.
- Antidepressant + Double-blind Placebo: Subjects received assigned oral, once daily antidepressant therapy (either escitalopram oxalate, sertraline hydrochloride, venlafaxine hydrochloride extended release, or duloxetine hydrochloride) plus oral, once daily, double-blind placebo (matching SPD489) for 8 weeks.
- Total: Total of all reporting groups
Arm/Group | Antidepressant + Double-blind SPD489 | Antidepressant + Double-blind Placebo | Total
Number analyzed (Participants) | 211 | 213 | 424
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42 (11.63) | 42.6 (11.41) | 42.3 (11.51)
Age, Customized [Count of Participants; unit: Participants]
  18-55 years | 181 | 184 | 365
  56-65 years | 30 | 29 | 59
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 141 | 143 | 284
  Male | 70 | 70 | 140

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score at 8 Weeks
Description: MADRS is a validated, 10-item rating scale with each item being scored on a scale from 0-6 with a total score ranging from 0-60. Lower scores indicate a decreased severity of depression.
Time Frame: 8 weeks
Population: Full Analysis Set: Subjects who took at least 1 dose of randomized investigational product and who had at least 1 valid primary efficacy measurement of the MADRS total score after the Augmentation Baseline Visit (Visit 8).
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Antidepressant + SPD489: Antidepressant + SPD489 (Lisdexamfetamine dimesylate): Antidepressant (either escitalopram oxalate, sertraline hydrochloride, venlafaxine hydrochloride extended release, or duloxetine hydrochloride) oral, once daily + SPD489 (optimized as a 20, 30, 50, or 70 mg dose, oral, once daily), for 8 weeks.
- Antidepressant + Placebo: Antidepressant + Placebo: Antidepressant (either escitalopram oxalate, sertraline hydrochloride, venlafaxine hydrochloride extended release, or duloxetine hydrochloride) oral, once daily + Placebo (oral, once daily) for 8 weeks.
Arm/Group | Antidepressant + SPD489 | Antidepressant + Placebo
Number analyzed (Participants) | 209 | 213
units on a scale | -7.3 [-8.6 to -6.0] | -6.8 [-8.1 to -5.5]
Statistical Analysis 1: Comparison: Antidepressant + SPD489 vs Antidepressant + Placebo; Test type: Superiority or Other; p = 0.583, Mixed-effects Model for Repeat Measures; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-2.3 to 1.3], Standard Error of Mean 0.92

2. Secondary Outcome: Mean Change From Baseline in Sheehan Disability Scale (SDS) Total Score at 8 Weeks
Description: Designed to evaluate the extent to which illness symptoms impact a subject's life in 3 areas: work/school, social, and family/home. Each area is scored on a scale from 0 (no impairment) to 10 (highly impaired) with a total score ranging from 0 (unimpaired) to 30 (highly impaired). Lower scores translate into less impairment.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Antidepressant + SPD489 | Antidepressant + Placebo
Number analyzed (Participants) | 209 | 213
units on a scale | -4.9 [-5.8 to -4.0] | -4.3 [-5.2 to -3.4]
Statistical Analysis 1: Comparison: Antidepressant + SPD489 vs Antidepressant + Placebo; Test type: Superiority or Other; p = 0.354, Mixed-effects Model for Repeat Measures; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-1.9 to 0.7], Standard Error of Mean 0.65

3. Secondary Outcome: Percentage of Participants Achieving a 25% Response on the MADRS
Description: The percentage of subjects who achieved a 25% response (i.e. ≥25% reduction in MADRS total score from the Lead-in Baseline, Visit 2).
Time Frame: Up to 8 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Antidepressant + SPD489 | Antidepressant + Placebo
Number analyzed (Participants) | 209 | 213
percentage of participants | 68.9 | 74.2

4. Secondary Outcome: Percentage of Participants Achieving a 50% Response on the MADRS
Description: The percentage of subjects who achieved a 50% response (i.e. ≥50% reduction in MADRS total score from the Lead-in Baseline, Visit 2).
Time Frame: Up to 8 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Antidepressant + SPD489 | Antidepressant + Placebo
Number analyzed (Participants) | 209 | 213
percentage of participants | 41.6 | 37.1

5. Secondary Outcome: Percent of Participants Achieving Remission on the MADRS
Description: MADRS remission was defined as a MADRS total score of ≤10.
Time Frame: Up to 8 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Antidepressant + SPD489 | Antidepressant + Placebo
Number analyzed (Participants) | 209 | 213
percentage of participants | 23.0 | 17.8

6. Secondary Outcome: Mean Change From Baseline Over Time in MADRS Total Score
Description: as for outcome 1
Time Frame: Up to 8 weeks
Population: Full Analysis Set: Subjects who took at least 1 dose of randomized investigational product and who had at least 1 valid primary efficacy measurement of MADRS total score after the Augmentation Baseline Visit (Visit 8). Sample size (n) of MADRS total score at each visit differed from sample size (N) of the FAS.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Antidepressant + SPD489 | Antidepressant + Placebo
Number analyzed (Participants) | 209 | 213
units on a scale
  Week 9 (Visit 9) | -2.9 [-3.9 to -2.0] | -2.1 [-3.0 to -1.1]
  Week 10 (Visit 10) | -4.4 [-5.5 to -3.3] | -4.3 [-5.4 to -3.2]
  Week 11 (Visit 11) | -5.9 [-7.1 to -4.7] | -5.0 [-6.2 to -3.8]
  Week 12 (Visit 12) | -6.3 [-7.6 to -5.1] | -5.3 [-6.5 to -4.1]
  Week 14 (Visit 13) | -6.9 [-8.2 to -5.5] | -6.4 [-7.7 to -5.1]
  Week 16 (Visit 14) | -7.3 [-8.6 to -6.0] | -6.8 [-8.1 to -5.5]

7. Secondary Outcome: Mean Change From Baseline in Abbreviated Brief Assessment of Cognition Affective Disorders (ABAC-A) Composite T-Scores
Description: The ABAC-A is a rater-administered series of activities designed to be sensitive to the critical cognitive deficits in affective disorders and schizophrenia. There are 6 subtests of the ABAC-A: List Learning (verbal memory); Digit Sequencing Task (working memory); Token Motor Task (motor speed); Verbal Fluency; Symbol Coding (attention and processing speed); and Tower of London Test (executive functions). The ABAC-A Composite T-score change from Augmentation Baseline Visit (Visit 8; Week 8) at Visit 14/Early Termination (ET) (Week 16/ET) was analyzed.
Time Frame: up to 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: t-score
Arm/Group | Antidepressant + SPD489 | Antidepressant + Placebo
Number analyzed (Participants) | 194 | 198
t-score | 3.0 [2.1 to 4.0] | 2.5 [1.5 to 3.5]

8. Secondary Outcome: Mean Change From Baseline in the Short Form-12 Health Survey V2 (SF-12V2)
Description: Total score ranges from 0 (lowest level of health) - 100 (highest level of health) on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability (i.e. a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability). Higher scores are associated with better quality of life.
Time Frame: Up to 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Antidepressant + SPD489 | Antidepressant + Placebo
Number analyzed (Participants) | 196 | 205
units on a scale
  Physical | 1.07 [0.04 to 2.10] | 0.90 [-0.11 to 1.91]
  Mental | 6.63 [5.03 to 8.23] | 5.16 [3.60 to 6.73]

9. Secondary Outcome: Mean Change in Sexual Functioning Questionnaire - 14 Item Scale (CSFQ-14) Total Score Male
Description: The CSFQ-14 is a short-form interview/questionnaire that measures illness- and medication-related changes in sexual functioning. A 5-point Likert scale is used ranging from 1 (never) to 5 (always). The CSFQ-14 total score can range from 14 to 70, with lower scores being associated with worsened sexual functioning.
Time Frame: Up to 8 weeks
Population: Full Analysis Set: Male subjects who took at least 1 dose of randomized investigational product and who had at least 1 valid primary efficacy measurement of the MADRS total score after the Augmentation Baseline Visit (Visit 8).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Antidepressant + SPD489 | Antidepressant + Placebo
Number analyzed (Participants) | 64 | 67
units on a scale | 2.1 (6.22) | 1.0 (6.02)

10. Secondary Outcome: Mean Change in Sexual Functioning Questionnaire - 14 Item Scale (CSFQ-14) Total Score Female
Description: as for outcome 9
Time Frame: Up to 8 weeks
Population: Full Analysis Set: Female subjects who took at least 1 dose of randomized investigational product and who had at least 1 valid primary efficacy measurement of the MADRS total score after the Augmentation Baseline Visit (Visit 8).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Antidepressant + SPD489 | Antidepressant + Placebo
Number analyzed (Participants) | 125 | 133
units on a scale | 3.0 (7.11) | 1.9 (5.82)

11. Secondary Outcome: Clinical Global Impressions - Global Improvement (CGI-I)
Description: Clinical Global Impression-Improvement (CGI-I) consists of a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved) or 2 (much improved) on the scale.
Time Frame: Up to 8 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Antidepressant + SPD489 | Antidepressant + Placebo
Number analyzed (Participants) | 209 | 213
percentage of participants
  Improved | 56.9 | 53.5
  Not Improved | 43.1 | 46.5
  Not Assessed | 0 | 0

12. Secondary Outcome: Mean Change From Baseline in the Multidimensional Assessment of Fatigue (MAF) Global Fatigue Index (GFI)
Description: MAF contains 16 items scored on a scale from 1 (not at all) to 10 (a great deal). Answers are converted to a Global Fatigue Index with total scores ranging from 1 (no fatigue) to 50 (severe fatigue). Lower scores indicate less fatigue.
Time Frame: Up to 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Antidepressant + SPD489 | Antidepressant + Placebo
Number analyzed (Participants) | 197 | 205
units on a scale | -6.6 (0.74) | -4.4 (0.73)

13. Secondary Outcome: Columbia Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS is a semi-structured interview that captures the occurence, severity, and frequency of suicide-related thoughts and behaviors during the assessment period. The interview includes definitions and suggested questions to solicit the type of information needed to determine if a suicide-related thought or behaviour occurred. The assessment is done by the nature of the responses, not by a numbered scale.
Time Frame: Up to 8 weeks
Population: Safety Analysis Set: All subjects who took at least 1 dose of randomized investigational product and who had at least 1 safety assessment (e.g., coming back for any visit, reporting of an adverse event [AE], or reporting the absence of AEs) after the Augmentation Baseline Visit (Visit 8).
Measure: Number; unit: percentage of participants
Arm/Group | Antidepressant + SPD489 | Antidepressant + Placebo
Number analyzed (Participants) | 211 | 213
percentage of participants
  ≥1 positive suicidal ideation | 9.0 | 9.4
  ≥1 suicidal attempt | 0 | 0.5

14. Secondary Outcome: Amphetamine Cessation Symptom Assessment (ACSA) - Total Aggregate Score
Description: ACSA scale has 16 symptom items rated on a scale from 0 (not at all) to 4 (extremely) with a possible total score range of 0 to 64. Higher scores indicate greater withdrawal symptom severity.
Time Frame: 8 weeks
Population: Safety Analysis Set: All subjects who took at least 1 dose of randomized investigational product and who had at least 1 safety assessment (e.g., coming back for any visit, reporting of an AE, or reporting the absence of AEs) after the Augmentation Baseline Visit (Visit 8).
Measure: Mean (Standard Deviation); unit: Score
Groups:
- Antidepressant + SPD489: Antidepressant + SPD489 (Lisdexamfetamine dimesylate): Antidepressant (either escitalopram oxalate, sertraline hydrochloride, venlafaxine hydrochloride extended release or duloxetine hydrochloride) oral, once daily + SPD489 (optimized as a 20, 30, 50, or 70 mg dose, oral, once daily), for 8 weeks.
Arm/Group | Antidepressant + SPD489 | Antidepressant + Placebo
Number analyzed (Participants) | 194 | 199
Score | 17.0 (10.80) | 17.2 (10.56)

ADVERSE EVENTS:
Groups:
- SPD489: Antidepressant + SPD489 (Lisdexamfetamine dimesylate ): Antidepressant (either escitalopram oxalate, sertraline hydrochloride, venlafaxine hydrochloride extended release or duloxetine hydrochloride) oral, once daily + SPD489 (oral, 20, 30, 50 or 70 mg, once daily) for 8 weeks
- Placebo: Antidepressant + Placebo: Antidepressant (either escitalopram oxalate, sertraline hydrochloride, venlafaxine hydrochloride extended release or duloxetine hydrochloride) oral, once daily + Placebo (oral, once daily) for 8 weeks
Arm/Group | SPD489 | Placebo
Serious Adverse Events (participants affected / at risk) | 1/211 | 1/213
Other Adverse Events (participants affected / at risk) | 72/211 | 46/213
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SPD489 (N=211) | Placebo (N=213)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Accelerated hypertension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SPD489 (N=211) | Placebo (N=213)
Dry mouth (Gastrointestinal disorders) | 25 (29) | 6 (6)
Nasopharyngitis (Infections and infestations) | 14 (14) | 19 (20)
Decreased appetite (Metabolism and nutrition disorders) | 13 (14) | 5 (5)
Headache (Nervous system disorders) | 25 (32) | 16 (22)
Insomnia (Psychiatric disorders) | 11 (14) | 7 (7)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 11 (16) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.